CLINICAL TRIAL: NCT02654483
Title: A Phase 2 Trial of Neurokinin-1 Receptor Antagonist for the Treatment of Itch in Epidermolysis Bullosa Patients
Brief Title: Neurokinin-1 Receptor Antagonist for the Treatment of Itch in EB Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jean Yuh Tang (Other)
Collaborators: Epidermolysis Bullosa Research Partnership (Other Government); Vyne Therapeutics Inc. (Industry)
Responsible Party: Sponsor-Investigator, Jean Yuh Tang, Associate Professor, Stanford University
Organization: Stanford University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 34182
Record Dates: First submitted 2016-01-11; First posted 2016-01-13 (Estimated); Results first posted 2019-07-02 (Actual); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Epidermolysis Bullosa; Pruritus
MeSH Terms: conditions — Epidermolysis Bullosa; Pruritus | interventions — serlopitant

STUDY DESIGN:
Intervention Model Description: Phase 2 investigator-initiated, randomized, double-blind, placebo-controlled, parallel-arm trial evaluating the comparative effect of serlopitant 5 mg by mouth daily versus placebo in treatment of chronic pruritus in pediatric and adult EB patients
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Research personnel not involved in this study was responsible for blinding. This was the only personnel with access to the code linking study drug bottle numbers to treatment (i.e. active or placebo). The code was broken when all data was captured and locked on an electronic data capture system.
Oversight: Data Monitoring Committee: No

ARMS (2):
- 5 mg VPD-737 (Experimental): 5 mg tablets of VPD-737 to be taken daily by mouth for 56 days
  Interventions: Drug: VPD-737
- Placebo (Placebo Comparator): Placebo tablets to be taken daily by mouth for 56 days
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: VPD-737 — VPD-737 inhibits the receptor neurokinin-1.
  Other Names: Serlopitant
  Arms: 5 mg VPD-737
Other: Placebo — Matching tablets to VPD-737 tablets without active drug
  Arms: Placebo

SUMMARY:
Our goal is to determine whether daily oral administration of VPD-737 (5 mg) is effective and safe in treating moderate to severe pruritus in patients with Epidermolysis Bullosa (EB).

DETAILED DESCRIPTION:
Itch is the most common complaint reported by patients with EB of all subtypes, and there is no current effective treatment. Itch often triggers scratching that creates new wounds and increases EB disease severity.

This study aims to target the physiological mechanisms of pruritus (itch) in patients with EB. Substance P is a major mediator of pruritus and binds to the receptor neurokinin-1 (NK1), which is expressed in the central nervous system and the skin.

VPD-737 (serlopitant), a novel drug that inhibits the NK1 receptor, has been shown to reduce severe itch in a previous study of 257 adult patients with chronic pruritus.

Each patient will be un-blinded individually after completing 3 months of study period.

All patients who complete the study will be offered a 2-month period on active drug. Patient who received active drug in the first period will be contacted and asked if they would like to continue on active drug for an additional 2 months.

Patients who received placebo in the first period will be contacted and asked if they would like to repeat the study on open label for 2 months.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Epidermolysis Bullosa (EB) and pruritus

Exclusion Criteria:

* Chronic liver or renal disease

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2016-08-31 (Actual); Primary Completion 2018-06-28 (Actual); Study Completion 2018-07-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean Tang, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chiou AS, Choi S, Barriga M, Dutt-Singkh Y, Solis DC, Nazaroff J, Bailey-Healy I, Li S, Shu K, Joing M, Kwon P, Tang JY. Phase 2 trial of a neurokinin-1 receptor antagonist for the treatment of chronic itch in patients with epidermolysis bullosa: A randomized clinical trial. J Am Acad Dermatol. 2020 Jun;82(6):1415-1421. doi: 10.1016/j.jaad.2019.09.014. Epub 2019 Sep 18. PMID 31541747
- See also: Phase 2 trial of a neurokinin-1 receptor antagonist for the treatment of chronic itch in patients with epidermolysis bullosa: A randomized clinical trial. — https://www-ncbi-nlm-nih-gov.laneproxy.stanford.edu/pubmed/31541747

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A 30-day washout period from prohibited medications (if applicable) is included prior to arm assignment.
  All patients who complete the double-blinded period will be offered a 2-month period on active drug.
Period: Double-blind
Arm/Group | 5 mg VPD-737 | Placebo
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0
Period: Open-label
Arm/Group | 5 mg VPD-737 | Placebo
Started (6 participants in total did not continue to the open-label period) | 5 (2 participants did not proceed to open-label arm) | 3 (4 participants did not continue to open-label arm)
Completed | 5 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All study participants
Groups:
- Total: Total of all reporting groups
Arm/Group | 5 mg VPD-737 | Placebo | Total
Number analyzed (Participants) | 7 | 7 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.6 (12.1) | 22.9 (8.0) | 25.2 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 3 | 4 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 5 | 5 | 10
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 6 | 3 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 3 | 4
Region of Enrollment [Number; unit: participants]
  United States | 7 | 7 | 14
NRS daily itch severity score [Mean (Standard Deviation); unit: score on a scale] — Mean daily itch score as measured by patient self-reports using a numeric rating scale (NRS) for itch severity and the Stanford EB itch questionnaire. NRS is included in the Stanford EB Itch survey. The NRS is comprised of one item and represents the numbers 0 ("no itch") to 10 ("worst imaginable itch").
  score on a scale | 6.1 (1.9) | 6.6 (1.0) | 6.6 (1.2)
NRS itch severity during bathing/dressing change [Mean (Standard Deviation); unit: score on a scale] — Mean itch score during bathing/dressing change as measured by patient self-reports using a numeric rating scale (NRS) for itch severity and the Stanford EB itch questionnaire. NRS is included in the Stanford EB Itch survey. The NRS is comprised of one item and represents the numbers 0 ("no itch") to 10 ("worst imaginable itch").
  score on a scale | 6.1 (1.9) | 6.2 (2.2) | 6.1 (1.9)
EB wound size [Mean (Standard Deviation); unit: mm^2] — Target wounds are identified and quantified at baseline using the Canfield image analysis system.
  mm^2 | 42.6 (65.8) | 25.0 (21.9) | 34.2 (48.3)

OUTCOME MEASURES:

1. Primary Outcome: Comparative Weekly Change in NRS Itch Score Over the 8-week Active Treatment Period
Description: Determine the efficacy of Serlopitant compared with placebo on reducing EB-associated daily itch score as measured by patient self-reports using a numeric rating scale (NRS) for itch severity.The NRS is comprised of one item and represents the numbers 0 ("no itch") to 10 ("worst imaginable itch"). Because itch is subjective and can vary day to day, nightly NRS scores were recorded in patients' Itch Diaries. NRS recorded by subject daily, from screening visit through the end of the study.
  This study was designed to detect differences between the two treatment groups. The primary endpoint was the comparative weekly change in Numeric Rating Scale (NRS) itch severity score from baseline over 8 weeks; derived from a linear mixed effects model which utilizes observations from both the treatment and placebo groups to generate an interaction term of interest. Itch severity changes from day to day and this model can more appropriately report trends in patients' itch severity with treatment.
Time Frame: Baseline and 8 weeks
Population: The relative effect of drug on the mean daily change in NRS itch severity score as compared to baseline is calculated and serves as the primary endpoint. Data is reported as point/week change (delta) in NRS itch score.
Measure: Mean (95% Confidence Interval); unit: score/week comparative change
Groups:
- 5 mg VPD-737: 7 subjects were treated with active drug
- Placebo: 7 subjects were treated with placebo
Arm/Group | 5 mg VPD-737 | Placebo
Number analyzed (Participants) | 7 | 7
score/week comparative change | -2 [-5 to 0] | -1 [-7 to 1]

2. Secondary Outcome: Wound Healing Determination
Description: Wound dimensions, including length, width, and area (in cm2), will be obtained using the Canfield system. Changes in dimensions between visits as well as changes in dimensions from baseline will be recorded. Overall mean % change from baseline is reported as the secondary endpoint.
Time Frame: Baseline and 8 weeks
Population: Eligible participants were: age 13 and older with a clinical diagnosis of EB and a Numeric Rating Scale (NRS) score for pruritus of ≥4 at baseline on average itch or itch during bathing or dressing in the past 24 hours. Patients were required to have itch symptoms lasting ≥6 weeks that did not respond well to the current standard of care.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | 5 mg VPD-737 | Placebo
Number analyzed (Participants) | 7 | 7
percentage change | 154.54 (227) | 38.39 (180)

3. Secondary Outcome: Change in Mean NRS Itch Score During Bathing/Dressing Changes
Description: Itch is exacerbated by activities such as dressing changes or bathing. NRS itch score during bathing or dressing in the past 24 hours were collected. Numeric rating scale (NRS) for itch severity is comprised of one item and represents the numbers 0 ("no itch") to 10 ("worst imaginable itch"). This study was designed to detect differences between the two treatment groups. This secondary endpoint was the comparative change in Numeric Rating Scale (NRS) itch severity score during bathing/dressing changes from baseline over 8 weeks as determined by application of a linear mixed effects model.
Time Frame: Baseline and 8 weeks
Population: The relative effect of drug on the mean change in NRS itch severity score during dressing changes as compared to baseline is calculated and serves as the secondary endpoint.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | 5 mg VPD-737 | Placebo
Number analyzed (Participants) | 7 | 7
score on a scale | -2.5 [-4 to 1] | -2 [-5 to 0]

ADVERSE EVENTS:
Time Frame: Up to 10 months; some patients did not proceed to the open-label arm immediately and were monitored for AEs during the period between arms.
Description: AE grading by severity based on judgement of investigators. Grade I = mild, Grade II = moderate, Grade III = severe. AEs were captured/followed at all study visits.
Groups:
- Double-blind, 5 mg VPD-737: 5 mg tablets of VPD-737 to be taken daily by mouth for 56 days
  VPD-737: VPD-737 inhibits the receptor neurokinin-1.
- Double-blind, Placebo: Placebo tablets to be taken daily by mouth for 56 days
  Placebo: Matching tablets to VPD-737 tablets without active drug
- Open-label, 5 mg VPD-737 - 5 mg VPD-737: 5 mg tablets of VPD-737 to be taken daily by mouth for 56 days, followed by a wash out period and, 5 mg tablets of VPD-737 to be taken daily by mouth for 2 months.
- Open-label, Placebo - 5 mg VPD-737: Placebo tablets to be taken daily by mouth for 56 days, followed by a wash out period and, 5 mg tablets of VPD-737 to be taken daily by mouth for 2 months.
Arm/Group | Double-blind, 5 mg VPD-737 | Double-blind, Placebo | Open-label, 5 mg VPD-737 - 5 mg VPD-737 | Open-label, Placebo - 5 mg VPD-737
All-Cause Mortality (participants affected / at risk) | 0/7 | 1/7 | 0/5 | 0/3
Serious Adverse Events (participants affected / at risk) | 1/7 | 1/7 | 0/5 | 0/3
Other Adverse Events (participants affected / at risk) | 6/7 | 7/7 | 2/5 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Double-blind, 5 mg VPD-737 (N=7) | Double-blind, Placebo (N=7) | Open-label, 5 mg VPD-737 - 5 mg VPD-737 (N=5) | Open-label, Placebo - 5 mg VPD-737 (N=3)
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
heart failure (Cardiac disorders) | 1 | 0 | 0 | 0
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
nephropathy (Renal and urinary disorders) | 0 | 1 | 0 | 0
hematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Double-blind, 5 mg VPD-737 (N=7) | Double-blind, Placebo (N=7) | Open-label, 5 mg VPD-737 - 5 mg VPD-737 (N=5) | Open-label, Placebo - 5 mg VPD-737 (N=3)
nausea (Gastrointestinal disorders) | 2 | 1 | 0 | 0
diarrhea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
otitis (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
headache (Nervous system disorders) | 1 | 1 | 0 | 1
somnolence (Nervous system disorders) | 0 | 1 | 0 | 0
dizziness (Nervous system disorders) | 1 | 1 | 0 | 0
infection (wound) (Infections and infestations) | 2 | 2 | 0 | 1
exacerbation of pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
flu-like symptoms (General disorders) | 1 | 0 | 0 | 0
cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
pain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 — unrelated to biopsy site
toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 0
infection (Infections and infestations) | 1 | 1 | 0 | 0 — bronchial
fever (General disorders) | 0 | 1 | 0 | 0
skin ulceration (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
upper respiratory infection (Infections and infestations) | 1 | 0 | 1 | 0
constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 1
dysesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 — formication
pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 — facial/jaw pain
dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2019-04-17): https://cdn.clinicaltrials.gov/large-docs/83/NCT02654483/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2017-01-09): https://cdn.clinicaltrials.gov/large-docs/83/NCT02654483/Prot_SAP_001.pdf